CLINICAL TRIAL: NCT02825602
Title: Vietnam Era Health Retrospective Observational Study
Acronym: VE-HEROeS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Veteran Affairs Office of Patient Care Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Victoria J. Davey PhD, MPH, Senior Investigator, Epidemiology Program, Veteran Affairs Office of Patient Care Services
Other Study IDs: 15-12
Record Dates: First submitted 2016-06-13; First posted 2016-07-07 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Aging; Combat Disorders
Keywords: Vietnam veteran; aging; health; War Injury; Conventional Warfare; Toxic Effect; Chemical
MeSH Terms: conditions — Combat Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Vietnam War Theater Veterans: Vietnam War Theater Veterans are defined for this protocol as those who served in the U.S. Armed Forces on the ground, in the air, or on the inland waters of Vietnam, Cambodia, and/or Laos between February 28, 1961 and May 7, 1975, inclusive. The investigators based this definition on legal dates of service set forth in 38 Code of Federal Regulations (CFR) 3.2 - Periods of war, but broadened the definition of sites of military service that constituted war zones based on written historical accounts and input from Vietnam Veterans.
- Blue Water Navy Vietnam Veterans: Blue Water Navy Veterans are defined as Veterans who served aboard deep-water naval vessels in waters offshore North or South Vietnam between February 28, 1961 and May 7, 1975 and who never served ashore or on inland waterways of Vietnam.
- Vietnam era Veterans: Vietnam era Veterans served in locations around the world OTHER than on the ground, in the air, or on the inland waters of Vietnam, Cambodia, and/or Laos or aboard deep-water naval vessels in waters offshore North or South Vietnam between February 28, 1961 and May 7, 1975.
- Non-military U.S. public: Non-military U.S. public are individuals who were born before 1958, never served in the U.S. military, and are age- and gender-matched (by the study investigators) to Vietnam War Theater Veterans.

SUMMARY:
The Vietnam Era Health Retrospective Observational Study (VE-HEROeS) is a national study on the health and well-being of Vietnam Veterans, including Blue Water Navy Veterans, as well as Veterans who served elsewhere during the Vietnam Era (1961-1975), and similarly aged U.S. residents who never served in the military. The investigators will invite approximately 43,000 Vietnam and Vietnam Era Veterans, and approximately 11,000 members of the general U.S. population to participate in VE-HEROeS. These individuals are scientifically selected to participate; the study is not able to accept volunteers.

All participants in VE-HEROeS will be asked to fill out a questionnaire on their military service, general health, age-related conditions, health care use, and the health experiences of their children and grandchildren. A smaller group will be asked to provide the investigators with access to some of their medical records. Topics of special focus for the study include cognition, hepatitis C infection, and neurologic conditions.

DETAILED DESCRIPTION:
It has been more than 40 years since the Vietnam War ended and there is little recent systematic knowledge of how Veterans of the Vietnam Era (1961-1975) have fared with regard to their overall health, lifestyle factors, and aging. This epidemiologic study, called the Vietnam Era Health Retrospective Observational Study (VE-HEROeS) will provide information about the health and well-being of Veterans of the Vietnam Era to Veterans and their families who have questions about the long-term health effects of service during the Vietnam War, to clinicians who care for Veterans and lack sufficient evidence to explain health conditions, and to the VA healthcare system in order to improve VA healthcare and anticipate future healthcare needs. The main objective of this study is to determine if the overall health of Veterans of the Vietnam War and Vietnam Era, with a special focus on neurologic conditions and hepatitis C infection, is different from that of their counterparts who did not serve in the military. Exploratory aims of the study are to determine if the investigators can obtain a sample of Blue Water Navy Vietnam Veterans (who served exclusively in deep coastal waters off of North or South Vietnam) and use the survey to describe their current health, and to determine the prevalence of Veterans who attribute health conditions of their descendants to their own military service, especially conditions potentially transmitted epigenetically. The study design is a survey, with hepatitis C and neurologic conditions validated by medical record review. The questionnaire includes both validated scales and new items about physical and mental health, exposures, and lifestyle. There are two versions of the questionnaire: one for Veterans of the Vietnam Era and one for those selected from the U.S. general population who have never served in the military. The questionnaires are as similar as possible, with the exception of questions about military service, exposures, or experiences that are either removed or modified in the non-Veteran questionnaire because they do not apply to this population.

ELIGIBILITY:
Inclusion Criteria:

* invited to participate through investigators' random sample selection process
* able to provide informed consent
* have a postal address in the U.S. or its territories

Exclusion Criteria:

* individuals who are incarcerated
* individuals who are unable to complete the survey even with assistance because of cognitive or physical limitations.

Min Age: 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans: We will obtain a stratified random sample of 45,067 Veterans from the Department of Veterans Affairs' United States Veterans Eligibility Trends & Statistics (USVETS) database which we believe to be the most complete database of U.S. military Veterans in existence. Stratification will be on period of service within the Vietnam era: 1961-1964 or 1965-1975. We will remove decedents and those without a current US postal address from the sample.
  U.S. public: The U.S. public general population comparison sample will be an age- and gender-matched sample of living non-Veteran members of the U.S. public born before 1958.
Sampling Method: Probability Sample
Enrollment: 24306 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03-31 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall Health | Past 4 weeks
  Overall health will be measured by the mean physical component summary score (PCS) and the mean mental component score (MCS) of the Short Form 8 (SF-8) compared across the four groups. Mean scores on the 8 health concepts measured by the SF-8 (physical functioning, role limitations due to physical functioning, bodily pain, general health, energy/fatigue, social functioning, role limitations due to emotional problems, and psychological distress/well being) will also be compared. Adjustments may be made for age, gender, and prevalent co-morbidities.

SECONDARY OUTCOMES:
Conditions of concern | Health history assessed at the time of survey (Day 1)
  The investigators will compare post-war prevalence of conditions that have been linked to Vietnam War service in other scientific studies of multiple designs: neurologic conditions ( Parkinson's disease, dementia, stroke, brain injury), Hepatitis C; hypertension, ischemic heart disease, Type II diabetes, peripheral neuropathy, various cancers, cirrhosis, alcohol and drug dependency.

OTHER OUTCOMES:
Self-identification of Blue Water Navy Vietnam Veterans | Navy service exclusively in the deep offshore waters of Vietnam between February 28, 1961 and May 7, 1975.
  The investigators will ask Blue Water Navy Veterans to define themselves by their response to a survey question, as no roster of these Veterans exists.
Health of offspring | Health history assessed at the time of survey (Day 1)
  We ask survey respondents to report 9 conditions of their children and grandchildren that may be transmitted epigenetically

CONTACTS AND LOCATIONS:
Overall Officials: Victoria J Davey, PhD, MPH, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- U.S. Department of Veterans Affairs/Epidemiology Program, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate data will be available to investigators in accordance with VA access policy.

REFERENCES:
- [Background] Health status of Vietnam veterans. II. Physical Health. The Centers for Disease Control Vietnam Experience Study. JAMA. 1988 May 13;259(18):2708-14. PMID 2833631
- [Background] Health status of Vietnam veterans. I. Psychosocial characteristics. The Centers for Disease Control Vietnam Experience Study. JAMA. 1988 May 13;259(18):2701-7. PMID 2833630
- [Background] Health status of Vietnam veterans. III. Reproductive outcomes and child health. The Centers for Disease Control Vietnam Experience Study. JAMA. 1988 May 13;259(18):2715-9. PMID 2833632
- [Background] Kulka RA, Schlenger WE, Fairbank JA, Hough RL, Jordan BK, Marmar CR, et al. Trauma and the Vietnam War Generation. New York: Brunner/Mazel Publishers; 1990
- [Background] Institute of Medicine (US) Committee to Review the Health Effects in Vietnam Veterans of Exposure to Herbicides. Veterans and Agent Orange: Health Effects of Herbicides Used in Vietnam. Washington (DC): National Academies Press (US); 1994. Available from http://www.ncbi.nlm.nih.gov/books/NBK236356/ PMID 25144022
- [Background] Dominitz JA, Boyko EJ, Koepsell TD, Heagerty PJ, Maynard C, Sporleder JL, Stenhouse A, Kling MA, Hrushesky W, Zeilman C, Sontag S, Shah N, Ona F, Anand B, Subik M, Imperiale TF, Nakhle S, Ho SB, Bini EJ, Lockhart B, Ahmad J, Sasaki A, van der Linden B, Toro D, Martinez-Souss J, Huilgol V, Eisen S, Young KA. Elevated prevalence of hepatitis C infection in users of United States veterans medical centers. Hepatology. 2005 Jan;41(1):88-96. doi: 10.1002/hep.20502. PMID 15619249
- [Background] Raymont V, Salazar AM, Krueger F, Grafman J. "Studying injured minds" - the Vietnam head injury study and 40 years of brain injury research. Front Neurol. 2011 Mar 28;2:15. doi: 10.3389/fneur.2011.00015. eCollection 2011. PMID 21625624
- [Background] Bullman TA, Kang HK. Posttraumatic stress disorder and the risk of traumatic deaths among Vietnam veterans. J Nerv Ment Dis. 1994 Nov;182(11):604-10. doi: 10.1097/00005053-199411000-00002. PMID 7964667
- [Background] Marmar CR, Schlenger W, Henn-Haase C, Qian M, Purchia E, Li M, Corry N, Williams CS, Ho CL, Horesh D, Karstoft KI, Shalev A, Kulka RA. Course of Posttraumatic Stress Disorder 40 Years After the Vietnam War: Findings From the National Vietnam Veterans Longitudinal Study. JAMA Psychiatry. 2015 Sep;72(9):875-81. doi: 10.1001/jamapsychiatry.2015.0803. PMID 26201054
- [Background] Manikkam M, Tracey R, Guerrero-Bosagna C, Skinner MK. Dioxin (TCDD) induces epigenetic transgenerational inheritance of adult onset disease and sperm epimutations. PLoS One. 2012;7(9):e46249. doi: 10.1371/journal.pone.0046249. Epub 2012 Sep 26. PMID 23049995
- [Background] The association of selected cancers with service in the US military in Vietnam. III. Hodgkin's disease, nasal cancer, nasopharyngeal cancer, and primary liver cancer. The Selected Cancers Cooperative Study Group. Arch Intern Med. 1990 Dec;150(12):2495-505. doi: 10.1001/archinte.150.12.2495. PMID 2244766
- [Background] The association of selected cancers with service in the US military in Vietnam. I. Non-Hodgkin's lymphoma. The Selected Cancers Cooperative Study Group. Arch Intern Med. 1990 Dec;150(12):2473-83. PMID 2244764
- [Background] The association of selected cancers with service in the US military in Vietnam. II. Soft-tissue and other sarcomas. The Selected Cancers Cooperative Study Group. Arch Intern Med. 1990 Dec;150(12):2485-92. PMID 2244765
- [Background] Kang HK, Cypel Y, Kilbourne AM, Magruder KM, Serpi T, Collins JF, Frayne SM, Furey J, Huang GD, Kimerling R, Reinhard MJ, Schumacher K, Spiro A 3rd. HealthViEWS: mortality study of female US Vietnam era veterans, 1965-2010. Am J Epidemiol. 2014 Mar 15;179(6):721-30. doi: 10.1093/aje/kwt319. Epub 2014 Jan 30. PMID 24488510
- [Background] Institute of Medicine (US) Committee on Blue Water Navy Vietnam Veterans and Agent Orange Exposure. Blue Water Navy Vietnam Veterans and Agent Orange Exposure. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK209599/ PMID 24983057
- [Derived] Blosnich JR, Hilgeman MM, Cypel YS, Akhtar FZ, Fried D, Ishii EK, Schneiderman A, Davey VJ. Potentially traumatic events and health among lesbian, gay, bisexual and heterosexual Vietnam veterans: Results from the Vietnam Era Health Retrospective Observational study. Psychol Trauma. 2022 May;14(4):568-577. doi: 10.1037/tra0001025. Epub 2021 Jun 17. PMID 34138613